CLINICAL TRIAL: NCT02057094
Title: Effect of Protein Supplementation on Lean Body Mass Recovery and Physiological Resilience Following Survive, Evade, Resist, Escape (SERE) School
Brief Title: Effects of Protein Supplementation on Lean Body Mass Recovery From Extreme Military Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 14-02H
Record Dates: First submitted 2013-12-05; First posted 2014-02-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2015-04

CONDITIONS: Military Operational Stress Reaction; Malnutrition (Calorie); Weight Loss; Muscle Wasting
MeSH Terms: conditions — Malnutrition; Weight Loss; Muscular Atrophy | interventions — Proteins; Whey

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Dining facility recovery feeding only, no supplemental protein consumed (an isoenergetic, carbohydrate supplement will be consumed by those assigned to the Control group)
  Interventions: Dietary Supplement: Protein, High-Protein, and Control
- Protein (Active Comparator): Consume dining facility food with:
  2, 20 g whey protein supplements daily (for ~27 days)
  1, 40 g casein protein supplement daily (for ~27 days)
  Interventions: Dietary Supplement: Protein, High-Protein, and Control
- High-Protein (Active Comparator): Consume dining facility food with:
  2, 40 g whey protein supplements daily (~27 days)
  1, 50 g casein protein supplement daily (~27 days)
  Interventions: Dietary Supplement: Protein, High-Protein, and Control

INTERVENTIONS:
Dietary Supplement: Protein, High-Protein, and Control
  Other Names: Whey and Casein protein; Carbohydrate-based control

SUMMARY:
The purpose of this study is to evaluate the physiological consequences of extreme military training and determine whether protein supplementation enhances recovery by promoting gains in lean body mass. This study will be conducted at the US Marine Survive, Evade, Resist, Escape (SERE) school at Camp Lejeune, North Carolina.

SERE school may be an ideal setting to assess nutritional interventions that promote recovery from severe military operational stress, and identify innate or experiential variables that may lead to increased levels of resilience in Warfighters. Our laboratory has recently demonstrated the detrimental effects and stressful nature of SERE. Heart rates and stress-related hormones increased dramatically, with concomitant reductions in circulating anabolic hormones. Additionally, SERE causes significant weight loss (15-20 lbs), which probably included lean body mass. The effects of severe operational stress induced by SERE, particularly the loss of lean mass, may degrade physical performance, increase injury risk, and compromise military readiness. Under controlled laboratory conditions, consuming high protein diets or supplemental high-quality protein promotes muscle protein retention, enhances muscle protein synthesis, and protects lean body mass in response to stress. Whether consuming supplemental protein promotes lean mass recovery and physiological resilience following a 'real-world' military stress has not been determined. Further, the level of supplemental protein necessary to optimize recovery from extreme military operational stress has not been elucidated.

Up to 90 US Marines will be enrolled in a 46-day double-blind, placebo-controlled trial. Using complex body composition measurements, kinetic modeling of human metabolism, blood sampling and cognitive and nutrition questionnaires, the consequences of SERE and the efficacy of protein recovery nutrition on lean mass accretion and Warfighter resilience will be assessed.

We hypothesize that consuming a specially formulated, high-quality supplemental protein ration item will speed recovery of lean body mass, physiological, and psychological resilience following extreme military operational stress.

ELIGIBILITY:
Inclusion Criteria:

* US Marines at least 18 years old, enrolled in US Marine SERE school

Exclusion Criteria:

* Self-reported allergies to dairy products

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in lean body mass following SERE and recovery nutrition | days 1-2, days 18-19, and days 45-46
  Days 1-2: baseline Days 18-19: completion of SERE training Days 45-46: completion of a 26 day recovery nutrition intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Pasiakos, Ph.D., Principal Investigator — USARIEM Military Nutrition Division
Locations (1):
- US Marine SERE School, Marine Corps Base Camp Lejeune, North Carolina, United States

REFERENCES:
- [Background] Berryman CE, Sepowitz JJ, McClung HL, Lieberman HR, Farina EK, McClung JP, Ferrando AA, Pasiakos SM. Supplementing an energy adequate, higher protein diet with protein does not enhance fat-free mass restoration after short-term severe negative energy balance. J Appl Physiol (1985). 2017 Jun 1;122(6):1485-1493. doi: 10.1152/japplphysiol.01039.2016. Epub 2017 Apr 6. PMID 28385919
- [Derived] Berryman CE, McClung HL, Sepowitz JJ, Gaffney-Stomberg E, Ferrando AA, McClung JP, Pasiakos SM. Testosterone status following short-term, severe energy deficit is associated with fat-free mass loss in U.S. Marines. Physiol Rep. 2022 Sep;10(18):e15461. doi: 10.14814/phy2.15461. PMID 36117330